CLINICAL TRIAL: NCT03656042
Title: A Open-label, No-treatment-controlled, Parallel, Pilot Phase Ⅱ Study to Evaluate the Efficacy and Safety/Tolerability Profiles of G-CSF in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: To Evaluate the Efficacy and Safety/Tolerability Profiles of G-CSF in Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 96-0272A-ASAD-061202
Record Dates: First submitted 2018-08-23; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2017-02

CONDITIONS: Alzheimer's Disease
Keywords: Dementia; Alzheimer's disease; Granulocyte-colony stimulating factor
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- G-CSF (Experimental): Subjects in the treatment group will receive Filgrastim (75mcg/0.3ml, NEUPOGEN®), 10 mic/kg/day, by sc, for 5 continuous days for the first week, rest for 11 weeks. Filgrastim will be given 12-weekly ( 12 weeks/cycle ) for 2 cycles.
  Interventions: Drug: Filgrastim (75mcg/0.3ml)
- No-treatment (No Intervention): No-treatment group is used to control evaluation bias and potential time effect.

INTERVENTIONS:
Drug: Filgrastim (75mcg/0.3ml) — Subjects who meet all eligible requirements for entry into the study will be randomized into one of the two treatment groups in 1:1 ratio as shown below:
  1. 10 microgram/kg/day, by sc, for 5 continuous days for the first week, rest for 11 weeks; repeat dosing regimen every 12-weekly (12 weeks / cycle) for 2 cycles
  2. Non-treatment
  Other Names: NEUPOGEN®
  Arms: G-CSF

SUMMARY:
With the enrichment of living environment and the progress of medicine, the scale of aging population has increased in many countries of the world. Alzheimer's disease (AD), the leading cause of dementia, counts for approximately 60% to 70% in dementia in aged population. AD is a well-known neurodegenerative disease and characterized by the formation of neurofibrillary tangles and deposition of amyloid in the brain. It also affects more than 12 million patients worldwide and puts a tremendous burden on family caregivers and causes high nursing home costs for society. So far, the mechanisms of AD have not been elucidated and currently no curable treatment exists. Thus, clinical trials concerning the treatment of AD are in urgent expectation.

Granulocyte-colony stimulating factor (G-CSF) is a growth factor that presents in human body in small quantity and is known to promote the blood cell proliferation and differentiation. Previous studies showed injection of G-CSF could help release hematopoietic stem cell (HSCs) from bone marrow to the peripheral blood, and then migrate to repair damaged areas, e.g. heart tissue and ischemia brain tissue. We have found that G-CSF triggering release of stem cells from bone marrow shows the potential as an effective reagent for treatment of AD by using two AD mouse models. The one was generated by injecting the brains of normal mice with amyloid and another was by using a strain of transgenic mice which naturally exhibit Alzheimer's disease-like neuronal apoptosis and memory loss. Subcutaneous administration of G-CSF into mice significantly rescued their cognitive/memory functions.

G-CSF has already been widely used in clinical practice, for example, neutropenia caused by chemotherapy in cancer and bone marrow transplantation. The new finding shows G-CSF can release HSCs from bone marrow and these cells not only can pass through the blood-brain barrier but can selectively migrate to the region of damaged brain to improve neurological recovery. Thus, we conduct this clinical trial to investigate the potential effect of G-CSF for the cognitive function of AD patients. If successful, G-CSF could open up a new window for AD treatment which is less invasive and more effective than the current therapies.

DETAILED DESCRIPTION:
This is a randomized open-label Phase 2 trial with parallel design using no-treatment group as control. Subjects in the treatment arm will receive subcutaneous G-CSF with the dosage of 10 microgram/kg/day, for 5 continuous days in the first week. The second dosage will be given in the 12 week. If subjects has received Donepezil already, the Donepezil will be concomitantly used in a stable dose (the same dose as pre-entering this study) during the study.

Background data and general medical history will be registered on the screening visit (Visit 1, started four weeks or less before Visit 2). Subjects fulfil the inclusion criteria 1) age between 50 to 85 years old; 2) those who were diagnosed as AD and the supporting evidences from the brain computed tomography or Magnetic Resonance Imaging scan within 12-months; 3) Mini-Mental State Examination scores of 10 to 26, and, 4) Clinical Dementia Rating score of 1 or 2. Subjects with clinically significant medical or neurological disorders, other than AD, that may affect cognition will be excluded Additional inclusion criteria included Modified Hachinski Ischemic score of ≤ 4, Hamilton Psychiatric Rating Scale for Depression score of ≤ 12and a reliable caregiver who is sufficiently familiar with the subject and is willing to provide the accurate data.

Participants will receive standard physical examination in all visits. Serum tests include complete blood count (CBC),total bilirubin, creatinine, blood urea nitrogen (BUN), uric acid, aspartate transaminase (AST), alanine transaminase (ALT), total protein, albumin, Vitamin B12, folate, T4, thyroid-stimulating hormone (TSH), HbA1c, rapid plasmin reagin (RPR)/Treponema pallidum haemagglutination (TPHA) will be also obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with age of at lease 50 years old and no more than 85 years old
2. Subject diagnosed of Alzheimer's disease; based on the criteria of The Diagnostic and Statistical Manual of Mental Disorders (DSM)-Ⅳ for dementia and those of National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Dementia and Related Disorder Association (NINCDS - ADRDA) and within 12-months CT/MRI brain scan supporting evidences.
3. Subject with Mini-Mental Examination (MMSE) scores of 12 to 26 (inclusive).
4. Subject with Clinical Dementia Rating (CDR) score of 1 (mild) or 2 moderate).
5. Subject with Modified Hachinski Ischemic score of 4.
6. Subject with a Hamilton Psychiatric Rating Scale for Depression score of 12.
7. Female subject with child-bearing potential agrees to take reliable contraceptive method during the participation of the study (Females with no child-bearing potential have to be surgically sterilized or at least 2 years after post-menopausal).
8. Subject and subject's legally acceptable representative have given written informed consent.
9. A reliable caregiver is sufficiently familiar with the subject (as determined by the investigator) and is willing to provide accurate data.

Exclusion Criteria:

1. Subject has underwent any of the following treatment modalities with the respective time frames:

   1. Anti-epileptic agents: Within 12 weeks of the screening visit,
   2. Narcotic: within 12 weeks of the screening visit,
   3. Immunosuppressants: within 12 weeks of the screening visit,
   4. Hypnotics: within 24 hours of the screening visit or the randomization visit,
   5. Lithium: within 2 weeks of the randomization visit,
   6. Succinylcholine-type muscle relaxants: within 2 weeks of the randomization visit,
   7. Drugs or treatments known to cause major organ system toxicity: within 42 weeks of the randomization visit,
   8. Tricyclic and tetracyclic anti-depressants: within 4 weeks of the screening visit,
   9. Antiparkinsonian: Within12 weeks of the screening visit (Not including dopaminergic agent or peripheral anticholinergic agent at stable dose for at least 4 weeks of randomization visit),
   10. Any medications for cognition enhancement: Within13 weeks of the screening visit(except for donepezil that has been maintained with a stable regimen for at least 12 weeks).
2. Subject is lactating, pregnant or plans to become pregnant,
3. Subject is cared primarily by nursing home,
4. Subject's AST or ALT is greater than 2 times of the upper limit or normal range.
5. Subject with diabetic history and with HbA1c > 8.5 %.
6. Subject with clinically significant medical or neurological disorders, other than AD, that may affect cognition (e.g., abnormal thyroid function tests, Vitamin B12 or folate deficiency, post-traumatic conditions Huntington's disease, Parkinson's disease, syphilis, probable/possible vascular dementia according to NINDS-AIREN criteria, active/uncontrolled seizure).
7. Subject with major psychiatric disorders.
8. Subject with spleen related disorders.
9. Subject with sickle cell disease.
10. Subject with myelodysplastic syndrome.
11. Subject with current diagnosis of acute stroke or history of acute stroke within 1 year.
12. Subject with allergy history to E. coli-derived proteins or G-CSF or donepezil.
13. Subject with cancer history and has received related therapy(ies) with in 2 years of entering this study.
14. Subject has participated other investigational study within 4 weeks of entering this study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale, Cognitive subscale - Chinese version (ADAS-Cog-C) | 24 weeks
  The total score ranges from 0 to 75 and the higher the score, the greater the impairment. ADAS-Cog-C has 11 items and each has its score range:
  Word Recall Task: maximum score = 10 Naming Task: maximum score = 5 Commands: maximum score = 5 Constructional Praxis: maximum score = 5 Ideational Praxis: maximum score = 5 Orientation: maximum score = 8 Word Recognition: maximum score = 12 Remembering Test Instructions: maximum score = 5 Spoken Language Ability: maximum score = 5 Word-Finding Difficulty: maximum score = 5 Comprehension: maximum score = 5 We measure the change from baseline in ADAS-Cog at 24-week visit.

SECONDARY OUTCOMES:
Mini-mental State Examination (MMSE) | Baseline, 12 weeks, 24 weeks and 48 weeks
  The Mini-Mental State Examination (MMSE) is a 30-point questionnaire.
  The score ranges are as follows:
  Orientation to time 5 Orientation to place 5 Registration 3 Attention and calculation 5 Recall 3 Language 2 Repetition 1 Complex commands 5
Clinical Dementia Rating Scale (CDR) | Baseline, 12 weeks, 24 weeks and 48 weeks
  The Clinical Dementia Rating Scale is a 5-point scale used to characterize six domains of cognitive and functional performance to Alzheimer disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care.
  In each domain, the severity degree of each symptom correspond to different rating score from 0(none) to 3(severe). The total score ranges from 0 to 18
AD Cooperative Study - Clinical Global Impression of change (ADCS-CGIC ) | Baseline, 12 weeks, 24 weeks and 48 weeks
  Interviewer scores the severity as follow:
  1. Not impaired / not present
  2. Borderline impairment
  3. Mild impairment
  4. Moderate impairment
  5. Marked impairment
  6. Severe impairment
  7. very severe
Lawton and Brody Scale for Instrumental Activities of Daily Living (IADL) | Baseline, 12 weeks, 24 weeks and 48 weeks
  The test measures eight realms of function through self report, which attempt to assess everyday functional competence in the elderly. Each item is rated either dichotomously (0 = less able, 1 = more able) or trichotomously (1 = unable, 2 = needs assistance, 3 = independent) and sum the eight responses. The summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men.
Neuropsychiatric Inventory (NPI) | Baseline, 12 weeks, 24 weeks and 48 weeks
  The NPI originally examined 12 sub-domains of behavioral functioning Each domain is scored for frequency, severity and associated caregiver distress.
  Frequency:Rarely,Sometimes,Often,Very often Severity:Mild,Moderate,Severe Caregiver Distress:0(not at all),1(minimally),2(mildly),3(moderately),4(severely),5(very severely or extremely). Total score will range from Less than 20(symptoms are mild),20-50(symptoms are moderate) to 50 or over(symptoms are severe)
Ten-point clock test (TPCT) | Baseline, 12 weeks, 24 weeks and 48 weeks
  One point is given for each of the following numbers that falls in its proper eighth of the circle relative to the number 12: 1.2, 4,5,7, 8, 10, and 11. One point is given each to a short hand pointing at the number eleven, and a long hand pointing at the number two. The total score ranges from 0 to 10.
CD34+ cell number for G-CSF treatment group | Baseline, 12 weeks, 24 weeks and 48 weeks
  G-CSF may promote mobilizing bone marrow CD34+ stem cells. We will compare the CD34+ cell number between treatment and control group at the baseline and follow up sequential change in the treatment group.
Trail making test (TMT)(Part A)) | Baseline, 12 weeks, 24 weeks and 48 weeks
  The Trail Making Test is a neuropsychological test of visual attention and task switching. Results for Trail making test A (Part A) is reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment. The average time is 29 seconds. If the subject uses more than 78 seconds, cognitive deficient is impressed.
Change from baseline in whole brain volume determined by MRI | Baseline, 24 weeks
  Change from baseline in whole brain volume determined by MRI. MRI examination will be performed within 7 days before the start at the start of first cycle (Visit 2) and week-24 visit (Visit 10), to compare the change of whole brain volume.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chuin Hsu, M.S., Principal Investigator — Chang Gung Memorial Hospital, Linkou medical center
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan R.o.c, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data sets including IPD that underlie results in a publication have not yet decided to be shared under the consideration of patient privacy.

REFERENCES:
- [Background] Alzheimer's Association. 2016 Alzheimer's disease facts and figures. Alzheimers Dement. 2016 Apr;12(4):459-509. doi: 10.1016/j.jalz.2016.03.001. PMID 27570871
- [Background] Scheltens P, Blennow K, Breteler MM, de Strooper B, Frisoni GB, Salloway S, Van der Flier WM. Alzheimer's disease. Lancet. 2016 Jul 30;388(10043):505-17. doi: 10.1016/S0140-6736(15)01124-1. Epub 2016 Feb 24. PMID 26921134
- [Background] Braak H, Del Tredici K. The preclinical phase of the pathological process underlying sporadic Alzheimer's disease. Brain. 2015 Oct;138(Pt 10):2814-33. doi: 10.1093/brain/awv236. Epub 2015 Aug 17. PMID 26283673
- [Background] Chartier-Harlin MC, Crawford F, Houlden H, Warren A, Hughes D, Fidani L, Goate A, Rossor M, Roques P, Hardy J, et al. Early-onset Alzheimer's disease caused by mutations at codon 717 of the beta-amyloid precursor protein gene. Nature. 1991 Oct 31;353(6347):844-6. doi: 10.1038/353844a0. PMID 1944558
- [Background] Tigue CC, McKoy JM, Evens AM, Trifilio SM, Tallman MS, Bennett CL. Granulocyte-colony stimulating factor administration to healthy individuals and persons with chronic neutropenia or cancer: an overview of safety considerations from the Research on Adverse Drug Events and Reports project. Bone Marrow Transplant. 2007 Aug;40(3):185-92. doi: 10.1038/sj.bmt.1705722. Epub 2007 Jun 11. PMID 17563736
- [Background] Yanqing Z, Yu-Min L, Jian Q, Bao-Guo X, Chuan-Zhen L. Fibronectin and neuroprotective effect of granulocyte colony-stimulating factor in focal cerebral ischemia. Brain Res. 2006 Jul 7;1098(1):161-9. doi: 10.1016/j.brainres.2006.02.140. Epub 2006 Jul 11. PMID 16814750
- [Background] Schneider A, Kruger C, Steigleder T, Weber D, Pitzer C, Laage R, Aronowski J, Maurer MH, Gassler N, Mier W, Hasselblatt M, Kollmar R, Schwab S, Sommer C, Bach A, Kuhn HG, Schabitz WR. The hematopoietic factor G-CSF is a neuronal ligand that counteracts programmed cell death and drives neurogenesis. J Clin Invest. 2005 Aug;115(8):2083-98. doi: 10.1172/JCI23559. Epub 2005 Jul 7. PMID 16007267
- [Background] Tsai KJ, Tsai YC, Shen CK. G-CSF rescues the memory impairment of animal models of Alzheimer's disease. J Exp Med. 2007 Jun 11;204(6):1273-80. doi: 10.1084/jem.20062481. Epub 2007 May 21. PMID 17517969
- [Background] Sanchez-Ramos J, Song S, Sava V, Catlow B, Lin X, Mori T, Cao C, Arendash GW. Granulocyte colony stimulating factor decreases brain amyloid burden and reverses cognitive impairment in Alzheimer's mice. Neuroscience. 2009 Sep 29;163(1):55-72. doi: 10.1016/j.neuroscience.2009.05.071. Epub 2009 Jun 14. PMID 19500657